CLINICAL TRIAL: NCT05790174
Title: Healthy Weight Development Among Children and Adolescents in the Central Denmark Region
Brief Title: Weight-loss Treatment Program in Children and Adolescents
Status: Active, not recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Healthy weight in children
Record Dates: First submitted 2023-02-14; First posted 2023-03-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-08

CONDITIONS: Childhood Obesity; Health Behavior; Weight Loss; Motivation
Keywords: Childhood obesity treatment
MeSH Terms: conditions — Pediatric Obesity; Health Behavior; Weight Loss

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: ROS "chubby and healthy" - a multidisciplinary family-based weight-loss treatment program — The weight-loss treatment program "ROS" is family-based and delivered by a multidisciplinary team of physicians, nurses, dieticians, and psychologists. The treatment is based on an individualized tailored plan made together with the family. The plan consists of dietary changes, more physical activity, regular weight checks, and motivational conversations. The program includes options of cooking classes, group session with a psychologist and participation in structured physical activity called "ROS sports" twice a week. Follow up visits are scheduled every 2-3 months at the different health care professionals.
Behavioral: Overweight Clinic for Children and Adolescents — The 'Overweight Clinic for Children and Adolescents' program at the municipal Health Center is based on the family-centered, multidisciplinary protocol developed by the Children's Obesity Clinic (TCOCT) at Holbæk Hospital. The intervention is individualized, informed by medical history and a structured questionnaire-based interview to identify behavioral and lifestyle changes needed to reduce the child's degree of overweight or obesity. The program consists of individual consultations every 6-8 weeks over approximately 12-18 months, with additional follow-up appointments as needed.
Behavioral: Family Nutrition Guidance — This treatment program is based on the Danish Health Authority's recommendations for lifestyle interventions. It follows a family-centered approach tailored to the family's everyday life and habits, focusing on sustainable changes in diet and physical activity. The program provides guidance on healthy eating, physical activity, and strategies for integrating these behaviors into daily routines.
  The program included the entire family and began with school-based consultations delivered by health nurses during the first three months, followed by additional sessions at the municipal Health Center when needed. Families were offered 4-6 consultations within the first six months and follow-up sessions twice a year.

SUMMARY:
The study will evaluate the effect of an existing municipality-based and hospital-based obesity treatment in children and adolescents in relation to weight loss and motivation. This is to ensure that children who have developed obesity have the possibility to obtain a healthier lifestyle, including a healthier body weight during their school years. This study will test whether an obesity treatment program designed for school children can reduce the degree of overweight in children and adolescents with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years old
* BMI SDS above the 90th percentile

Exclusion Criteria:

* Reached a BMI SDS below the 75th percentile
* Attained 19 years of age

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists of children and adolescents with overweight or obesity primarily living in Viborg, Skive, and Holstebro municipalities. Participants were offered either municipality-based treatment or a specialized hospital-based program. Municipality-based programs were delivered at local schools or health centers by health nurses or dietitians. The hospital-based program, offered by the Central Denmark Region, required referral from a general practitioner, school health nurse, or community-based physician.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in BMI during weight-loss program of childhood overweight and obesity | December 2022 - February 2026
  The primary objective is to investigate the changes in BMI z-score among children and adolescents with overweight or obesity who participated in a municipality-based or hospital-based weight-loss program, and whether existing characteristics of the child and parents at baseline modify this association. In addition we also want to characterize those who do not respond to treatment either because they gain or regain BMI z-score, or drop-out of the weight-loss program.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fogh M, Ostergaard JN, Jorgensen RM, Rossell EL, Eg M, Maindal HT, Toft G, Stovring H, Bruun JM. Long-Term Effect of a Hospital-Based Intervention Program on BMI Trajectories in Danish Children and Adolescents With Overweight and Obesity: A 6-Year Follow-Up. Clin Obes. 2026 Feb;16(1):e70052. doi: 10.1111/cob.70052. Epub 2025 Nov 2. PMID 41177529